CLINICAL TRIAL: NCT07270887
Title: The Long-term Effect of Remote Ischemic Conditioning on Main Organs in ASVCD Patients With Very High Risks (RICMO-ASCVD): a Prospective, Blinded Endpoint, Multi-center, Cohort Study
Brief Title: The Long-term Effect of Remote Ischemic Conditioning on Main Organs in ASVCD Patients With Very High Risks
Status: Recruiting | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Other Study IDs: Y (2025) 394
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: ASCVD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RIC group: The patients will receive treatment with RIC (5 cycles of cuff inflation for 5 minutes and deflation for 5 minutes to the bilateral upper limbs to 200 mmHg, twice daily) for 1 year as an adjunct to guideline-based treatment
  Interventions: Device: remote ischemic conditioning
- Control group: The patients will only receive guideline-based treatment

INTERVENTIONS:
Device: remote ischemic conditioning — 5 cycles of cuff inflation for 5 minutes and deflation for 5 minutes to the bilateral upper limbs to 200 mmHg
  Groups: RIC group

SUMMARY:
Atherosclerotic cardiovascular disease (ASCVD) is a group of disorders sharing atherosclerosis as a common pathological basis, primarily affecting the heart, brain, kidneys, and other peripheral arteries, leading to clinical syndromes characterized mainly by arterial ischemia. It has become the group of diseases with the highest morbidity and mortality rates worldwide. Patients with very high-risk ASCVD face an even greater risk of recurrence. Previous studies have discovered that remote ischemic conditioning (RIC) has protective effects on major organs such as the heart, brain, and kidneys. Given the cardiorenal and cerebrovascular protective effects of RIC, the invesitgators believe that long-term remote ischemic conditioning is a promising approach to preventing the recurrence of ASCVD events. Based on this hypothesis, the investigators have designed a prospective, multicenter cohort study with blinded outcome assessment to investigate the protective effects of long-term remote ischemic conditioning in very high-risk ASCVD populations.

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years
* Two or more prior major ASCVD events; OR one documented major ASCVD event with two or more of the following risk factors
* signed informed consent

Note： Definition of Major ASCVD Events:

A. Acute coronary syndrome within the past year. B. History of myocardial infarction (not part of a new acute coronary syndrome episode).

C. Ischemic stroke or history of ischemic stroke. D. Symptomatic peripheral artery disease, defined as intermittent claudication with an ankle-brachial index (ABI) < 0.85, or prior limb revascularization or amputation.

Risk factors:

1. Age ≥65 y
2. Heterozygous familial hypercholesterolemia
3. History of prior coronary artery bypass surgery or percutaneous coronary intervention outside of the major
4. ASCVD event(s)
5. Diabetes mellitus
6. Hypertension
7. CKD (eGFR 15-59 mL/min/1.73 m2)
8. Current smoking
9. Persistently elevated LDL-C (LDL-C ≥100 mg/dL [≥2.6 mmol/L]) despite maximally tolerated statin therapy and ezetimibe
10. History of congestive HF

Exclusion Criteria:

* Presence of severe neurological deficit (mRS score ≥ 3)
* Uncontrolled severe hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg despite medication)
* Subclavian artery stenosis ≥ 50% or presence of subclavian steal syndrome
* Severe hematological disorders or significant coagulation abnormalities
* Contraindications to remote ischemic conditioning, such as severe soft tissue injury, fracture, or vascular injury in the upper limbs, or peripheral vascular disease in the distal upper limbs
* Severe comorbid conditions with a life expectancy of less than 1 year
* Participation in another clinical trial within the past 3 months or ongoing participation
* Any other circumstances deemed by the investigator as unsuitable for participation in this clinical study.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: very high-risk ASCVD populations
Sampling Method: Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Composite Endpoint Events | 1 year
  including cardiovascular events, stroke, vascular death, and deterioration of renal function.

SECONDARY OUTCOMES:
Number of participants with no-fatal cardiovascular events | 1 year
Number of participants with no-fatal stroke | 1 year
Number of participants with no-fatal deterioration of renal function | 1 year
Change of renal function | 1 year
  renal function was meausred by serum urea nitrogen and creatinine
Change of blood pressure | 1 year
Changes in serological indicators such as blood glucose, blood lipids, and glycated hemoglobin (HbA1c) | 1 year
  Changes in the following serological indicators will be assessed and reported as separate outcome measures:
  Blood glucose (in mmol/L or mg/dL)
  Blood lipids [specify component, e.g., LDL-C, in mmol/L or mg/dL]
  Glycated hemoglobin (HbA1c) (in %)
Number of participants with new onset diabetes | 1 year
Occurence of vascular death | 1 year
Barthel Index (BI) scores | 1 year
  BI ranges from 0-100, higher scores meaning a better outcome.
Death due to all causes | 1 year

OTHER OUTCOMES:
Changes in cerebral small vessel disease burden (CSVD) | 1 year
  The total CSVD score is calculated by the following four neuroimaging features on MRI: lacunes, white matter hyperintensities, cerebral microbleeds and perivascular spaces (PVS). The score ranges from 0-4, with high score meaning heavier burden.
Changes in cognitive function measured by MoCA and MMSE | 1 year
  The Montreal Cognitive Assessment (MoCA) (score range: 0-30) and The Mini-Mental State Examination (MMSE) (score range: 0-30), with higher score meaning better cognitive function
Depressive symptoms measured by the Patient Health Questionnaire-9 (PHQ-9) | 1 year
  range from 0-27, higher score meaning worse symptoms
Anxiety symptoms measured by the Generalized Anxiety Disorder-7 (GAD-7) | 1 year
  range from 0-21, higher score meaning worse symptoms
Changes in cerebral autoregulation | 1 year
  cerebral autoregulation is measured by using TCD and Transfer Function Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China